CLINICAL TRIAL: NCT01911806
Title: Effectiveness of Back Care Pillow in Addition to Physical Therapy in Chronic Non-specific Low Back Pain Treatment
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Bundit Prommanon, school of physical therapy,Faculty of associated medical science,Khon Kaen University, Khon Kaen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MRG555S021
Record Dates: First submitted 2013-03-30; First posted 2013-07-30 (Estimated); Last update posted 2014-08-26 (Estimated); Status verified 2014-08

CONDITIONS: Chronic Nonspecific Low Back Pain
Keywords: Back care pillow; chronic non-specific low back pain; randomized controlled trial

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Back care pillow & standard physical therapy treatment (Experimental): standard physical therapy treatment for 6 sessions of treatment, each around 30 minutes, during a period of 2 weeks & back care pillow use during the day for 2 weeks
  Interventions: Device: Back care pillow; Procedure: standard physical therapy treatment
- standard physical therapy treatment (Active Comparator): standard physical therapy treatment for 6 sessions of treatment, each around 30 minutes, during a period of 2 weeks
  Interventions: Procedure: standard physical therapy treatment

INTERVENTIONS:
Device: Back care pillow — back care pillow is specific size by age groups of standard deviation of the lumbar spinal curvature, in 20-29 years was 51.68 ± 6.94 degrees, in 30-39 years was 59.67 ± 7.02 degrees, in 40-49 years was 63.66 ± 7.62 degrees, in 50-59 years was 65.75 ± 10.85 degrees and in 60-69 years was 64.19 ± 9.69 degrees
  Arms: Back care pillow & standard physical therapy treatment
Procedure: standard physical therapy treatment — standard physical therapy treatment are ultrasound therapy and hot pack

SUMMARY:
This study aim to investigate the effects of back care pillow, in adjective with standard physical therapy treatment for chronic non-specific low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Males or females
* Age 20 - 69 years old.
* Patients who have daily routine in so long bending of sitting or standing position at least 2 hours per day
* Patients with low back pain who have pain for more than 3 months
* Patients have pain at lower back without refer to leg
* Patients have moderate to severe pain of numerical rating scale (pain score ≥ 4)

Exclusion Criteria:

* Pregnant patients
* Underlying systematic or visceral disease, and specific condition such as neoplasm, ankylosing spondylitis, previous low back surgery
* Patients have Quada equine syndrome
* Patients with nerve root symptoms (neurological deficit)

  1. Patient have refer pain to leg area of same dermatome is problem.
  2. Abnormal reflex of lower extremity.
  3. Muscle weakness of area myotome is problem.

Ages: 20 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2013-03; Primary Completion 2013-07 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Pain Scores on the Numerical rating scale | three months

SECONDARY OUTCOMES:
Scale of lumbar range of motion measure by Modified - Modified Schober Test | three months

OTHER OUTCOMES:
Roland-Morris Disability Questionnaires (RMDQ) | three months

CONTACTS AND LOCATIONS:
Locations (1):
- School of physical therapy,Faculty of associated medical science,Khon Kaen University, Khon Kaen, Changwat Khon Kaen, Thailand